CLINICAL TRIAL: NCT06203080
Title: The Efficacy and Safety of an Intravaginal Acetic Acid Thermoreversible Gel on Chinese Women of Reproductive Age Compared With Nonoxinol Gel: A Multi-central Phase II, Triple-blind, Randomized Trial
Brief Title: The Contraceptive Efficacy and Safety of an Intravaginal Acetic Acid Thermoreversible Gel on Chinese Women.
Acronym: contraception
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Research Institute for Family Planning, China (Other Government)
Collaborators: Shanghai Jinxiang Latex Products Co. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NRIFP2023027
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Contraceptive Device; Complications
Keywords: contraception, STD
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): An acetic acid thermoreversible gel developed by Shanghai Jinxiang Latex Products Co. will be allocated to the intervention group.
  Interventions: Drug: ancetate gel
- Controlled group (Active Comparator): Nonoxinol gel produced by China Pharmaceutical University Pharmacy Co., Ltd will be allocated to the cotrolled group.
  Interventions: Drug: nonoxinol gel

INTERVENTIONS:
Drug: ancetate gel — An acetic acid thermoreversible gel produced by Shanghai Jinxiang Latex Products Co. will be utilized for the intervention. Each product weighs 4.85 g and contains 54.45 mg of poloxamer 407-acetic acid. The investigators will stockpile the product and distribute a total of 72 doses on the first day, at the end of the second month, and at the end of the fourth month of follow-up, respectively, after concealing the product's name. Participants will receive instructions to apply the medication transvaginally, one dose at a time, during each instance of sexual activity.
  Arms: Intervention group
Drug: nonoxinol gel — The nonoxinol gel produced by China Pharmaceutical University Pharmacy Co., Ltd will be utilized for the intervention. Each product weighs 5 g and contains 50 mg of N-9. The investigators will stockpile the product and distribute a total of 72 doses on the first day, at the end of the second month, and at the end of the fourth month of follow-up, respectively, after concealing the product's name. Participants will receive instructions to apply the medication transvaginally, one dose at a time, during each instance of sexual activity.
  Arms: Controlled group

SUMMARY:
The study aims to explore the efficacy and safety of an intravaginal acetic acid thermoreversible gel in Chinese women of reproductive age, comparing it with nonoxinol gel by assessing the six-month Pearl Index and the incidence of any side effects.

DETAILED DESCRIPTION:
Despite significant increases in the availability and effectiveness of contraceptives globally, there are few female-led devices that combine contraception and STI prevention. Previous studies suggested that acetic acid thermoreversible gel, a female targeted contraception, can regulate intravaginal ph, killing sperm and STI pathogens and protecting intravaginal probiotics. Therefore, we have developed a contraceptive gel containing 11.23 mg/g of poloxamer 407-acetic acid. To determine its contraceptive effectiveness and safety compared with the widely used nonoxinol gel, we will recruit about 240 reproductive-aged women in four centers in China and randomly allocate into two groups. During a six-month follow-up, we will compared their pregnant rates and incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 1) Aged between 20 and 45 years old;
* 2) Regular menstrual cycles (cycle length 25-35 days, menstruation lasting up to 7 days);
* 3) Have a history of pregnancy with the current partner at least once;
* 4) Currently engaging in regular sexual activity and planning to do so in the next six months (at least once a week);
* 5) Have not used hormonal contraceptive methods in the past 3 months;
* 6) Normal menstrual cycles have resumed after the removal of an intrauterine device;
* 7) Normal menstrual cycles have resumed after a previous miscarriage;
* 8) Breastfeeding women with normal menstrual cycles resumed;
* 9) No apparent gynecological abnormalities confirmed through examination, and normal cervical cytology (Pap smear grade I according to the Bethesda system);
* 10) Reliance on the investigational drug as the sole contraceptive method during the study period;
* 11) Willing to participate in this study, adhere to required follow-up visits, and voluntarily sign the informed consent form.

Exclusion Criteria:

* 1) Amenorrhoea for more than 1 month, suspected pregnancy;
* 2) Moderate to severe erosive changes in the cervix;
* 3) Vaginal cleanliness grade III or above;
* 4) Trichomonas, fungal vaginitis, and bacterial vaginosis, among other conditions, have not been cured;
* 5) Uterine prolapse of degree II or above and severe protrusion of the anterior and posterior vaginal walls;
* 6) Unexplained vaginal bleeding;
* 7) Genital tract deformities;
* 8) Malignant tumors of the genital tract;
* 9) Moderate or severe urinary incontinence;
* 10) Recurrent urinary tract infections;
* 11) History of allergy to acetic acid and/or nonoxinol.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Failure rate | Six months
  Pregnancy due to contraceptive failure under correct use and pregnancy due to incorrect and or discontinuous use will be respectively observed for six months for both groups.
Pregnancy rate during three months | Three months
  A cumulative incidence will be calculated according to the number of pregnancies during the first three months.
Pregnancy rate during six months | Six months
  A cumulative incidence will be calculated according to the number of pregnancies during the whole six months.
Termination rate during three months | Three months
  The termination due to any complications will be observed respectively in both groups during the first three months.
Termination rate during six months | Six months
  The termination due to any complications will be observed respectively in both groups during the whole six months.

SECONDARY OUTCOMES:
Complaint of adverse reactions | Six months
  Complaint rates of various adverse reactions (allergy/leucorrhoea/local irritation) during different follow-up time.
Biochemical index | Six months
  Biochemical index will be recorded respectively at the beginning of the follow-up and at the end of the follow-up through blood routine, urinalysis and liver function test.
Adherence use | Six months
  Adherence use will be evaluated during the follow-up respectively at the end of the first two weeks, two months, four months and six months through checking the number of used drugs packages and unused drugs.
Concomitant drugs | Six months
  Concomitant drugs will be recorded during the follow-up respectively at the end of the first two weeks, two months, four months and six months through the questionnaire.
Vaginal internal environment | Six months
  Vaginal microbiota examination will be used during the follow-up respectively at the end of the first two weeks, two months, four months and six months by professional physicians to evaluate the participant's vaginal internal environment whether is suitable for continuation of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Kaiyan Pei, MD, Principal Investigator — National Research Institute for Family Planning
Locations (4):
- China (4):
  - Beijing Shijitan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Central Hospital of Gynecology Obstetrics, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No